CLINICAL TRIAL: NCT06558890
Title: A Study on the Efficacy and Mechanism of Targeted Cerebellar Transcranial Electrical Stimulation for the Treatment of Refractory Temporal Lobe Epilepsy: A Single-center, Observational Study.
Brief Title: Transcranial Electrical Stimulation Targeting the Cerebellum for the Treatment of Refractory Temporal Lobe Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20232387
Record Dates: First submitted 2024-08-01; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-04

CONDITIONS: Transcranial Electrical Stimulation; Temporal Lobe Epilepsy; Magnetic Resonance Imaging; Electroencephalogram
MeSH Terms: conditions — Epilepsy, Temporal Lobe | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Alternating Current Stimulation Intervention (Experimental): Patients with refractory TLE recruited for the study will undergo a 6-week treatment with the tACS (transcranial alternating current stimulation) protocol, which involves a 2mA current at 10Hz for 20 minutes on both sides. The treatment schedule is 5 days of treatment followed by 2 days of rest, and then another 5 days of treatment, with a weekly reinforcement treatment, for a total of 14 sessions.
  Interventions: Device: Transcranial Alternating Current Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Transcranial Alternating Current Stimulation

SUMMARY:
Study the therapeutic effect and potential neural mechanisms of transcranial electrical stimulation targeting the cerebellum for the treatment of refractory temporal lobe epilepsy through MRI and EEG.

DETAILED DESCRIPTION:
This study is a single-center, observational study.This study applies transcranial alternating current stimulation to the cerebellum of patients with refractory temporal lobe epilepsy.For the recruited patients with refractory TLE (Temporal Lobe Epilepsy), they will undergo a 6-week treatment with tACS (transcranial alternating current stimulation) protocol (2mA, 10Hz, 20 minutes per side), following a schedule of treatment for 5 days - rest for 2 days - treatment for another 5 days, and then a reinforcement treatment once a week, completing a total of 14 treatments.Before treatment, at week 10, and at week 14, the frequency of epileptic seizures and the QOLIE-31 questionnaire scores will be recorded and assessed for the patients. EEG data and near-infrared spectroscopy (NIRS) brain functional imaging data will be collected before treatment and after two consecutive weeks of treatment. Magnetic resonance imaging (MRI) data will be acquired before treatment, after two consecutive weeks of treatment, and after six weeks of intensified treatment. Appropriate image processing methods and EEG processing methods will be utilized to analyze the changes in brain networks following tACS treatment, in order to explore the impact of tACS on the neural mechanisms of refractory temporal lobe epilepsy (TLE).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old;
2. Diagnosed with refractory temporal lobe epilepsy as defined by the International League Against Epilepsy (ILAE) (failure to achieve seizure-free status after adequate trials of two appropriate antiepileptic drugs);
3. Duration of epilepsy is at least 2 years, with a seizure frequency of at least 2 times per 4 weeks in the three months before enrollment;
4. Taking two or more antiepileptic drugs, and continuing the same medication treatment plan during the trial period;
5. Capable of cooperating to complete the treatment and related examination items;
6. The patient and family members fully understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Scalp skin damage (including skin diseases or damage in the area where electrodes are applied);
2. Psychogenic epilepsy or pseudo-epilepsy;
3. Concurrent severe infections, cerebrovascular diseases, malignant tumors, or other diseases with severe dysfunction of major organs such as the heart, liver, and kidneys, or with mental disorders;
4. Presence of any implanted devices or instruments (such as cardiac pacemakers, deep brain stimulators, cochlear implants, and vagus nerve stimulators, etc.);
5. History of head trauma or other brain-related diseases;
6. Pregnant or breastfeeding women;
7. Participation in other clinical trials at the same time;
8. Changes in medication treatment plan during baseline, treatment, or follow-up period;
9. Withdrawal of informed consent by the patient or family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Compared to baseline, the reduction rate of epileptic seizure frequency | baseline, 10 weeks,14 weeks after treatment
  ((post-treatment - baseline) / baseline).

SECONDARY OUTCOMES:
Quality of Life in Epilepsy-31 (QOLIE-31) Questionnaire | baseline, 10 weeks,14 weeks after treatment
  The scoring method for the QOLIE-31 Questionnaire involves several key steps, as follows:1.Initial Score Calculation： the raw scores for each item on the scale can be converted to a range of 0 to 100；2.Weighted Scoring：the transformed scores are multiplied by their respective weights；3.Total Score Calculation:all the weighted scores are added together to obtain the total score. Total Score=(Emotional Symptoms Score×25+Psychological Function Score×25+Social Function Score×20+Life Domains Score×17+Additional Items Score×13)/5 In the QOLIE-31 scoring system, a higher score indicates a better quality of life for individuals with epilepsy.
MRI measures | baseline，2weeks，14weeks after treatment
  This study primarily applied resting-state blood oxygen level dependent functional magnetic resonance imaging (BOLD) and magnetic resonance diffusion tensor imaging (DTI) techniques to evaluate the changes in functional connectivity of the cerebellum in healthy subjects and patients before and after two weeks of transcranial electrical stimulation (TES) treatment, as well as the changes in the cerebellar cortical white matter fiber bundles two months after treatment. ALFF and ReHo analyses can reveal the characteristics of local neural activity in the brain during the resting state, and abnormal brain regions can serve as regions of interest (ROIs) for subsequent functional connectivity analysis. Additionally, the flow of cerebrospinal fluid (CSF) can be measured to reflect the functional state of the glymphatic system, which can be used to assess the therapeutic effects and the impact on lymphatic drainage function.
electroencephalogram(EEG) | baseline，2weeks after treatment
  The changes in EEG will constitute secondary research outcomes. EEG can evaluate the changes in brain functional connectivity in patients before and after transcranial electrical stimulation (TES) treatment. In addition, the alterations in the power spectrum of each frequency band, including delta, alpha, beta, theta, low gamma, and high gamma, will also be measured before and after TES treatment.
Near-Infrared Spectroscopy (NIRS) Brain Functional Imaging | baseline，2weeks after treatment
  Near-Infrared Spectroscopy (NIRS) Brain Functional Imaging can assess the changes in brain function of patients before and after transcranial electrical stimulation (TES) treatment.Changes in brain functional connectivity as measured by near-infrared spectroscopy (fNIRS) imaging before and after transcranial electrical stimulation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wen, Study Chair — The First Affiliated Hospital of Air Force Medicial University
Locations (1):
- Xijing Hospital of Air Force Military Medical University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devinsky O, Vezzani A, O'Brien TJ, Jette N, Scheffer IE, de Curtis M, Perucca P. Epilepsy. Nat Rev Dis Primers. 2018 May 3;4:18024. doi: 10.1038/nrdp.2018.24. PMID 29722352
- [Background] Zoghi M, O'Brien TJ, Kwan P, Cook MJ, Galea M, Jaberzadeh S. Cathodal transcranial direct-current stimulation for treatment of drug-resistant temporal lobe epilepsy: A pilot randomized controlled trial. Epilepsia Open. 2016 Oct 17;1(3-4):130-135. doi: 10.1002/epi4.12020. eCollection 2016 Dec. PMID 29588936
- [Background] Theodore WH, Fisher RS. Brain stimulation for epilepsy. Lancet Neurol. 2004 Feb;3(2):111-8. doi: 10.1016/s1474-4422(03)00664-1. PMID 14747003
- [Background] Tergau F, Naumann U, Paulus W, Steinhoff BJ. Low-frequency repetitive transcranial magnetic stimulation improves intractable epilepsy. Lancet. 1999 Jun 26;353(9171):2209. doi: 10.1016/S0140-6736(99)01301-X. No abstract available. PMID 10392988
- [Background] Chen R, Spencer DC, Weston J, Nolan SJ. Transcranial magnetic stimulation for the treatment of epilepsy. Cochrane Database Syst Rev. 2016 Aug 11;(8):CD011025. doi: 10.1002/14651858.CD011025.pub2. PMID 27513825
- [Background] Liu A, Voroslakos M, Kronberg G, Henin S, Krause MR, Huang Y, Opitz A, Mehta A, Pack CC, Krekelberg B, Berenyi A, Parra LC, Melloni L, Devinsky O, Buzsaki G. Immediate neurophysiological effects of transcranial electrical stimulation. Nat Commun. 2018 Nov 30;9(1):5092. doi: 10.1038/s41467-018-07233-7. PMID 30504921
- [Background] Fregni F, Thome-Souza S, Nitsche MA, Freedman SD, Valente KD, Pascual-Leone A. A controlled clinical trial of cathodal DC polarization in patients with refractory epilepsy. Epilepsia. 2006 Feb;47(2):335-42. doi: 10.1111/j.1528-1167.2006.00426.x. PMID 16499758
- [Background] Antal A, Boros K, Poreisz C, Chaieb L, Terney D, Paulus W. Comparatively weak after-effects of transcranial alternating current stimulation (tACS) on cortical excitability in humans. Brain Stimul. 2008 Apr;1(2):97-105. doi: 10.1016/j.brs.2007.10.001. Epub 2007 Dec 3. PMID 20633376
- [Background] San-Juan D, Espinoza-Lopez DA, Vazquez-Gregorio R, Trenado C, Aragon MF, Perez-Perez D, Hernandez-Ruiz A, Anschel DJ. A pilot randomized controlled clinical trial of Transcranial Alternating Current Stimulation in patients with multifocal pharmaco-resistant epilepsy. Epilepsy Behav. 2022 May;130:108676. doi: 10.1016/j.yebeh.2022.108676. Epub 2022 Mar 30. PMID 35366528
- [Background] San-Juan D, Sarmiento CI, Hernandez-Ruiz A, Elizondo-Zepeda E, Santos-Vazquez G, Reyes-Acevedo G, Zuniga-Gazcon H, Zamora-Jarquin CM. Transcranial Alternating Current Stimulation: A Potential Risk for Genetic Generalized Epilepsy Patients (Study Case). Front Neurol. 2016 Nov 28;7:213. doi: 10.3389/fneur.2016.00213. eCollection 2016. PMID 27965623
- [Background] Mogul DJ, van Drongelen W. Electrical control of epilepsy. Annu Rev Biomed Eng. 2014 Jul 11;16:483-504. doi: 10.1146/annurev-bioeng-071813-104720. PMID 25014790
- [Background] Tavakoli AV, Yun K. Transcranial Alternating Current Stimulation (tACS) Mechanisms and Protocols. Front Cell Neurosci. 2017 Sep 1;11:214. doi: 10.3389/fncel.2017.00214. eCollection 2017. PMID 28928634
- [Background] Elyamany O, Leicht G, Herrmann CS, Mulert C. Transcranial alternating current stimulation (tACS): from basic mechanisms towards first applications in psychiatry. Eur Arch Psychiatry Clin Neurosci. 2021 Feb;271(1):135-156. doi: 10.1007/s00406-020-01209-9. Epub 2020 Nov 19. PMID 33211157
- [Background] Berenyi A, Belluscio M, Mao D, Buzsaki G. Closed-loop control of epilepsy by transcranial electrical stimulation. Science. 2012 Aug 10;337(6095):735-7. doi: 10.1126/science.1223154. PMID 22879515
- [Background] Streng ML, Krook-Magnuson E. The cerebellum and epilepsy. Epilepsy Behav. 2021 Aug;121(Pt B):106909. doi: 10.1016/j.yebeh.2020.106909. Epub 2020 Feb 5. PMID 32035793